CLINICAL TRIAL: NCT07002437
Title: Intermittent Hypoxia-Induced Motor Plasticity in Sub-Acute Spinal Cord Injury
Brief Title: Hypoxia Pathways for Early Recovery After Spinal Cord Injury
Acronym: HyPER-FLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202500467
Record Dates: First submitted 2025-05-02; First posted 2025-06-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Spinal Cord Injury; Intermittent Hypoxia; breathing; subacute; respiratory; acute intermittent hypoxia; hypoxia
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham (Sham Comparator): Participants will complete a baseline testing session, 6 sessions of sham intervention (5, 3-minute episodes of 21% O2, 2-minute intervals), and post-test assessments 1-day and 1-week after the last intervention.
  Interventions: Other: Sham AIH
- AIHH (Experimental): Participants will complete a baseline testing session, 6 sessions of acute intermittent hypercapnic hypoxia (AIHH) intervention (15, 1-minute episodes of 9-13% O2 + 4-5% CO2, 1.5-minute intervals), and post-test assessments 1-day and 1-week after the last intervention.
  Interventions: Other: Acute Intermittent Hypercapnic-Hypoxia (AIHH)
- aAIH (Experimental): Participants will complete a baseline testing session, 6 sessions of augmented acute intermittent hypoxia (aAIH) intervention (3, 5-minute episodes of 9-13% O2, 3-minute intervals), and post-test assessments 1-day and 1-week after the last intervention.
  Interventions: Other: Augmented Acute Intermittent Hypoxia (aAIH)

INTERVENTIONS:
Other: Augmented Acute Intermittent Hypoxia (aAIH) — aAIH (augmented acute intermittent hypoxia) consists of 3, 5-minute episodes of low oxygen (9-13% O2), interspersed with 3-min room air intervals.
  Each study participant will complete 6 sessions of augmented AIH (aAIH), which consists of 3, 5-minute exposures. Each exposure involves a 5-minute hypoxic episode (9-13% inspired O2), with a 3-min interval of room air breathing (21% O2). Gas mixtures will be delivered via Douglas bags (pre-filled with desired gas mixture) that are coupled to a non-rebreathing valve and facemask. A manual-control valve allows seamless gas mixture switching. Participant safety will be continuously monitored in real-time using non-invasive sensors and LabChart software. For instance, inspired and expired concentrations of O2 will be monitored by continuous recordings of arterial O2 saturation and end-tidal gas, respectively. Furthermore, vital signs (respiratory rate, tidal volume, heart rate, and blood pressure) will be continuously monitored.
  Arms: aAIH
Other: Acute Intermittent Hypercapnic-Hypoxia (AIHH) — AIHH consists of 1-min episodes of low oxygen (9% O2) and elevated carbon dioxide (5% CO2), interspersed with 1.5 min room air.
  Each participant will complete 6 sessions of AIHH exposure, which consists of 15, 1-minute hypercapnic hypoxic episodes (4-5% inspired CO2, 9-13% inspired O2), with 1.5-minute intervals of room air breathing (21% O2). Gas mixtures will be delivered in the same manner described for AIH intervention. Participant safety will be continuously monitored in real-time using LabChart software. For instance, inspired and expired concentrations of CO2 and O2 will be monitored by continuous recordings of arterial O2 saturation and end-tidal gas, respectively. Furthermore, vital signs (respiratory rate, heart rate, and blood pressure) will be monitored.
  Arms: AIHH
Other: Sham AIH — Six sessions of sham AIH with episodes of normal room air (21% O2).
  Sham experiments will use methods identical to AIH/AIHH protocols except that normoxic gas (21% inspired O2) will be delivered. Since the timing and intervals vary with each protocol, the sham will use a distinct protocol involving 5, 3-min episodes with 2 min intervals between each episode. The valve on the non-rebreathing mask will be turned to deliver these episodes, but 21% O2 will be delivered throughout.
  Arms: Sham

SUMMARY:
Spinal cord injury (SCI) disrupts neural pathways to respiratory motor neurons, diminishing breathing capacity and airway defense (e.g., cough). Indeed, respiratory impairment is a leading cause of infection, re-hospitalization and death after SCI. There is a critical need for new strategies to restore breathing ability and airway defense in people with SCI. Acute intermittent hypoxia (AIH) - repetitive exposure to brief episodes of low inspired oxygen - is a promising strategy to restore breathing capacity by promoting spinal neuroplasticity. Exciting outcomes in >12 SCI trials completed to date demonstrate that AIH improves human respiratory and limb function. Unfortunately, ~40% of individuals exhibit minimal response to AIH, making it essential to 1) optimize AIH protocols to maximize functional benefits; and 2) identify genetic biomarkers distinguishing those most/least likely to benefit from AIH-based treatments.

The purpose of the pilot study, to be conducted in a small sample of participants with sub-acute SCI (2 weeks to 6 months post injury), is to preliminarily compare the effects of two intermittent hypoxia protocols. Since AIH-induced plasticity may be induced via serotonin or adenosine-driven mechanisms and these pathways compete and inhibit each other, each protocol favors a distinct mechanistic pathway. Our long-term objective is to test the hypothesis that a longer duration (i.e., augmented) hypoxia protocol, favoring adenosine mechanisms, enhances respiratory motor plasticity more than an AIH protocol targeting serotonin mechanisms (low O2 + CO2) in people with sub-acute SCI. Since an individual's genetics can influence the response to rehabilitation, we are also investigating how certain genes are related to breathing changes after these treatments.

Data acquired through this pilot study will be used to inform a larger, more definitive clinical trial and will contribute to estimations of the magnitude and direction of effects.

DETAILED DESCRIPTION:
The specific focus of this pilot study is to obtain preliminary data to inform a larger, more definitive clinical trial. The long-term objective of this line of work is to test the hypothesis that an acute intermittent hypoxia protocol (3, 5 min episodes, 9-13% FiO2; augmented AIH (aAIH)) favoring adenosine mechanisms, enhances respiratory motor plasticity more than an AIH protocol targeting serotonin mechanisms (1 min 9% FiO2 + CO2) in people with sub-acute SCI. Since an individual's genetics can influence the response to rehabilitation, investigators are also collecting preliminary data regarding how certain genes are related to breathing changes after these treatments.

Data acquired through this pilot study will be used to estimate the magnitude and direction of effects.

This line of research will inform AIH protocol optimization to enhance the clinical effects of AIH treatments designed to improve rehabilitation outcomes.

The following Aims will be addressed:

Aim 1: To preliminarily test the hypothesis that augmented acute intermittent hypoxia (aAIH) is a more potent stimulus to induce respiratory motor plasticity than AIHH (low oxygen with hypercapnia) in people with sub-acute SCI.

The investigators predict that 6 sessions of aAIH (3, 5-minute episodes of 9-13% O2; 3-minute intervals) will elicit greater respiratory motor plasticity than AIHH (15, 1-minute episodes of 9-13% O2 with 4-5% CO2; 1.5-minute intervals) or Sham (5, 3-minute episodes of 21% O2) in individuals with SCI, 2 weeks to 6 months post injury.

The primary outcomes include maximum pressure generation and cough function 1-day and 1-week post-intervention. Secondary, exploratory outcomes will be biceps (elbow flexion) force output.

Aim 2: To obtain preliminary data regarding the association between dysfunctional genetic variants, linked with molecules necessary for AIH-induced respiratory motor plasticity, and the magnitude of response (change in primary outcomes) in response to aAIH or AIHH in individuals with sub-acute SCI.

The investigators predict that individuals with dysfunctional single nucleotide polymorphisms (SNPs) associated with pro-plasticity genes have blunted responses to aAIH and/or AIHH treatments.

* Augmented Acute intermittent hypoxia (aAIH): This intervention will involve breathing low-oxygen air through a facemask that covers the nose and mouth. Participants will be asked to breathe the low-oxygen air for 3 periods (about 5 minutes each period). A mask will be secured and adjusted to the face and the participant will be able to breathe naturally and normally. Between the ~ 5 minute periods of lower oxygen, the participant will breathe higher oxygen levels that are 'normal' or consistent with room air for about 3 minutes. Heart rate, blood oxygen saturation, and blood pressure will be monitored. The gas mixture will be adjusted if a participant's blood oxygen saturation drops below 80%.
* Acute intermittent hypercapnic hypoxia, lower oxygen with CO2 (AIHH): This intervention delivery using the facemask will be identical to the aAIH described above, except that lower oxygen will be combined with higher carbon dioxide air. For this intervention, the participant will be asked to breathe the low oxygen air with higher carbon dioxide air for 15 periods (~1 minute each). Between periods of breathing this gas mixture through the facemask, the participant will breathe higher oxygen levels that are normal for ~1.5 minutes. Heart rate, blood oxygen saturation, and blood pressure will be monitored. The gas mixture will be adjusted if a participant's blood oxygen saturation drops below 80%.
* Sham/Placebo: This intervention will be identical to the two procedures described above, except that normal-oxygen, normal-carbon dioxide air (same as room air) will be delivered through the facemask for 5 periods (~3 minutes each). Heart rate, blood oxygen saturation, and blood pressure will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18-70 years of age
2. Sub-acute incomplete SCI 2 weeks to 6 months after injury, at or below C1-T6 Incomplete SCI based on residual sensory and motor function below the level of the injury or injury classification of B, C, D at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI.

   -OR- Sub-acute complete SCI 2 weeks to 6 months after injury at or below C4-T6 Complete SCI based on the absence of residual sensory or motor function below the level of injury or injury classification of A at initial screening according to the American Spinal Injury Association Impairment Classification and the International Standards for the Neurological Classification of SCI.
3. Medically stable with physician clearance
4. SCI due to non-progressive etiology

Exclusion Criteria:

1. Current diagnosis of an additional neurologic condition such as Multiple Sclerosis, Parkinson disease, stroke, or brain injury
2. Severe illness or infection, including non-healing decubitus ulcers, untreated bladder or urinary tract infections, cardiovascular disease, lung disease, active heterotopic ossification, or uncontrolled hypertension
3. Severe neuropathic pain
4. Known pregnancy
5. Severe uncontrolled autonomic dysreflexia
6. Currently hospitalized in an acute care hospital

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Inspiratory Pressure | Baseline, 1-day, and 1-week following intervention
  Maximal inspiratory pressure is a non-invasive measure of the maximal force achieved when breathing in against an occluded airway.
Change in Maximal Expiratory Pressure | Baseline, 1-day, and 1-week following intervention
  Maximal expiratory pressure is a non-invasive measure of the maximal force achieved when breathing out against an occluded airway.
Change in Cough Function | Baseline, 1-day, and 1-week following intervention
  Cough function will be measured by non-invasive tests of cough volume acceleration during a maximal cough.

SECONDARY OUTCOMES:
Change in Muscle Strength | Baseline, 1-day, and 1-week following intervention
  Change in muscle strength will be measured using a non-invasive force dynamometer.

OTHER OUTCOMES:
Association between dysfunctional genetic variants necessary for AIH-induced respiratory motor plasticity with magnitude of response to AIH or AIHH interventions. | Once, at baseline.
  Genetic variants will be collected using a small saliva sample (2-5 mL) for genetic analysis to gain preliminary evidence regarding the effect of inter-individual genetic differences on response to AIH-based treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Fox, PT, DPT, MHS, PhD, Principal Investigator — University of Florida & Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No